CLINICAL TRIAL: NCT04199585
Title: Interventional, Randomized, Double-blind, Sequential-group, Placebo-controlled, Single-ascending Oral Dose Study Investigating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Lu AF95245 and Open-label Crossover Study to Investigate Intra-subject Variability, Effect of Food on Lu AF95245, and Metabolic Profile of [14C]-Lu AF95245 in Healthy Young Men
Brief Title: Safety and Tolerability of Lu AF95245 in Healthy Young Men
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: new safety data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18193A
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Cohort A: sequential, cohort B parallel
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: single-ascending oral dose (Experimental): Cohorts A1 to A6, single ascending dose, with 9 subjects in each cohort, sequential
  Interventions: Drug: Lu AF95245; Drug: Placebo
- Cohort B: (fasting/fed conditions) (Experimental): Groups B1, B2, and B3, with 4 subjects in each group and the groups will be running in parallel.
  B1: fed-fasting-fasting condition (spiked dosage)
  B2: fasting-fed-fasting condition (spiked dosage)
  B3: fasting-fasting-fed condition
  Interventions: Drug: Lu AF95245; Drug: Lu AF95245 14C radiolabelled spiked dosage

INTERVENTIONS:
Drug: Lu AF95245 — solution, single dose, orally
Drug: Lu AF95245 14C radiolabelled spiked dosage — solution, single dose, orally
  Arms: Cohort B: (fasting/fed conditions)
Drug: Placebo — solution, single dose, orally
  Arms: Cohort A: single-ascending oral dose

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of Lu AF95245 and what the body does to Lu AF95245 after swallowing single doses of the drug

DETAILED DESCRIPTION:
The study is divided in two parts, Part A and Part B:

Part A: interventional, randomized, double-blind, sequential-group, placebo-controlled, single-ascending oral dose study in healthy young men.

Part A will consist of up to 6 cohorts (Cohorts A1 to A6) with 9 subjects in each cohort. In each cohort, the subjects will be randomised to receive a single oral dose of Lu AF95245 or placebo (ratio 6:3)

Part B: interventional, randomized, open-label, three-period crossover study to investigate intra-subject variability, effect of food and mass balance and metabolic profile in healthy young men. Part B will be initiated when a anticipated therapeutically relevant dose confirmed to be safe and well-tolerated has been identified in Part A; this dose will be used in Part B. Part B is divided into 3 dosing periods and subjects will be randomised to 1 of 3 groups (Groups B1, B2, and B3) with 4 subjects in each group and the groups will be running in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young, non-smoking men with a body mass index (BMI) ≥18.5 kg/m2 and ≤30 kg/m2 at the Screening Visit.

Exclusion Criteria:

* The subject has any concurrent disorder that may affect the particular target or absorption, distribution, or elimination of the IMP.

Other in- and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | From baseline to Day 14
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, ECG parameters and physical examination)
AUC(0-inf) Lu AF95245 | From 0 to 96 hours
  Area under the plasma concentration time curve from zero to infinity
Cmax Lu AF95245 | From 0 to 96 hours
  Maximum observed plasma concentration
CL/F Lu AF95245 | From 0 to 96 hours
  Oral clearance for Lu AF95245 in plasma
Total recovery of the administered dose (% of dose in urine and faeces) | From 0 to Day 14
  Excretion of labelled Lu AF95245 in urine and faeces

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- QPS Netherlands BV, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided